CLINICAL TRIAL: NCT04858737
Title: Prevention of Depression in the Workplace Through a Personalized Intervention Based on Risk Algorithms, ICTs and Decision Support Systems: Randomized Controlled Trial
Brief Title: Personalized Prevention of Depression in the Workplace (e-pD-Work)
Acronym: e-pD-Work
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Mediterranean Institute for the Advance of Biotechnology and Health Research (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Institute of Biomedical Research in Málaga (IBIMA) (Unknown); Andalusian Regional Ministry of Health (Other Government); European Regional Development Fund (Other); University of Malaga (Other)
Responsible Party: Principal Investigator, Juan Ángel Bellón, PhD, Medicine, Andalusian Health Service
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PI18/01307
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Depression
Keywords: Depression; Primary prevention; Randomized controlled trial; m-Health; App; Workers
MeSH Terms: conditions — Depression; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-predicD-Work intervention (Experimental): In this arm, worker participants will receive an online personalized intervention to prevent depression based on ICTs, risk predictive algorithms and decision support systems (DSS).
  Interventions: Behavioral: e-predictD-Work intervention
- m-Health control (Active Comparator): In this arm, worker participants will continue receiving the usual care from their health providers. In addition, they will use an App with the same appearance as the e-predictD-Work App but it will only send weekly short messages about stress and general health that will be extracted from brochures and websites of official agencies.
  Interventions: Other: Brief psychoeducational messages

INTERVENTIONS:
Behavioral: e-predictD-Work intervention — The intervention is based on validated risk algorithms to predict depression and includes: 1) Mobile applications as main user's interface; 2) a DSS that helps worker participants to develop their own personalized plans to prevent (PPP) depression; 3) nine intervention modules (the core of the system) including activities to prevent depression, to be proposed by the DSS and chosen by the participants. The intervention is biopsychosocial and multi-component, including the following modules: physical exercise, improve sleep, expand relationships, solve problems, improve communication, assertiveness, decision making, manage thoughts and reduce work stress. Worker participants will implement the recommendations and the tool will monitor these actions, offering feedback to improve their PPP at 6 and 12 months.
  Arms: e-predicD-Work intervention
Other: Brief psychoeducational messages — The intervention consists of an App that weekly send short messages about stress and general health that will be extracted from brochures and websites of official agencies.
  Arms: m-Health control

SUMMARY:
The main goal is to design, develop and evaluate a personalized intervention to prevent depression in the workplace, based on Information and Communication Technologies (ICTs), predictive risk algorithms and decision support systems (DSS) for employed workers. The specific goals are: 1) to design and develop a DSS, called e-predictD-Work-DSS to elaborate personalized plans to prevent depression and its monitoring in the employed working population; 2) to design and develop an ICT solution that integrates the DSS on the web, a mobile application (App), the predictD risk algorithm, different intervention modules (including a work stress management module) and a monitoring-feedback system; 3) to evaluate the usability, adherence, acceptability and satisfaction of employed working population with the e-pD-Work intervention; 4) to evaluate the effectiveness of the e-pD-Work intervention to reduce the incidence of major depression, depression and anxiety symptoms, the probability of major depression next year and to improve quality of life; 5) to evaluate the cost-effectiveness and cost-utility of the e-pD-Work intervention to prevent depression.

Methods: This a randomized, double-blind, controlled trial with two parallel arms (e-pD-Work vs active m-Health control) and 12 months follow-up. A total of 3,160 depression-free workers, aged between 18 and 55 years old will be recruited in Spain and randomly assigned to one of the two groups in a 1:1 ratio considering a stratification of age (18-29, 30-39, 40-49, 50-55 years) and sex similar to the Spanish population. Participants, interviewers and statisticians will be blinded to participants' allocation. The e-pD-Work intervention is self-guided, has a biopsychosocial approach and is multi-component (9 modules: physical exercise, improve sleep, expand relationships, solve problems, improve communication, assertiveness, decision making, manage thoughts and reduce work stress). The e-pD-Work intervention will be implemented in the smartphone of the workers and pivot on an already validated risk predictive algorithm and a DSS that helps workers to develop their own personalized depression prevention plans. Primary outcome will be the rate of major depression measured by CIDI. As secondary outcomes: depressive and anxiety symptomatology measured by PHQ-9 and GAD-7 respectively, the risk probability of depression measured by the predictD risk algorithm, quality of life measured by SF-12 and EuroQol, and cost-effectiveness and cost-utility.

ELIGIBILITY:
Inclusion Criteria:

* Have a paid employement
* PHQ-9 <10 at baseline

Exclusion Criteria:

* Not have a smartphone and internet for personal use
* Sick leave for more than 1 month
* Unable to speak Spanish
* Documented terminal illness
* Documented cognitive impairment
* Documented serious mental illness (psychosis, bipolar, addictions, etc.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1054 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of major depression measured by the Composite International Diagnostic Interview (CIDI) | 12 months
  Composite International Diagnostic Interview (CIDI) is a structured diagnostic interview that provides current diagnoses of major depression according to DSM

SECONDARY OUTCOMES:
Depressive symptoms measured by the Patient Health Questionnaire-9 (PHQ-9) | 12 months
  The Patient Health Questionnaire-9 (PHQ-9) measures symptoms of depression through 9 items, each of which is scored 0 ('not at all') to 3 ('nearly every day'). Low scores are equivalent to less symptoms of depression, the scale range is 0 to 27 (9 items).
Anxious symptoms measured by the General Anxiety Questionnaire (GAD-7) | 12 months
  The General Anxiety Questionnaire (GAD-7) measures generalized anxiety disorder through 7 items, each of which is scored 0 ('not at all') to 3 ('nearly every day'). Low scores are equivalent to less symptoms of anxiety, the scale range is 0 to 21 (7 items).
Probability of depression measured by the Spanish predictD risk algorithm | 12 months
  The Spanish predictD risk algorithm reports a probability of suffering depression in the next 12 months measured by 13 risk factors. Scores range from 0% to 100%.
Quality of life measured by SF-12 | 12 months
  The 12-item Short Form (SF-12) measures quality of life related to physical health and quality of life related to mental health. Scores on the scales range from 0 to 100. Higher scores are equivalent to better health-related quality of life.
Satisfaction with paid work measured by an adapted version of the Job Content Instrument | 12 months
  The Job Content Instrument measures psychological demands, decision latitude, social support, physical demands, and job insecurity with a total of seven items. The first four are distributed on a 4-point Likert scale ranging from 'Often to Almost never / never), one of them is distributed on a dichotomous scale (yes / no), and the latter on a 4-point Likert scale ranging from 'Not at all to A lot'.
Acceptability and satisfaction with the interventions (e-predictD-Work intervention and m-Health control) measured by e-Health Impact Questionnaire | 12 months
  The e-Health Impact Questionnaire (e-HIQ) assesses the effects of websites containing health information. The e-HIQ questionnaire consists of two independently administered and scored parts. In the first part items represent general attitudes towards using the internet to access health information. In the second part items measure a person's ease with using online information, particularly emphasising a person's openness to learning and gaining support from other peoples experiences. Both parts of the questionnaire have a five point response category for all items ranging from 'Strongly disagree to Strongly agree'.
Cost-effectiveness | 12 months
  It will be conducted from two perspectives: (1) a societal perspective and (2) a National Health System perspective. We will calculate incremental cost-effectiveness ratio (ICER) using the incremental cost (difference in costs between arms) divided by incremental effectiveness (difference in the number of diagnoses of major depression between arms).
Cost-utility | 12 months
  It will be conducted from two perspectives: (1) a societal perspective and (2) a National Health System perspective. We will calculate incremental cost-effectiveness ratio (ICER) using the incremental cost (difference in costs between arms) divided by incremental QALYs (difference in QALYs between arms). Quality-adjusted life years (QALYs) will be measured using the EuroQol five questionnaire (EuroQol-5D).
Subgroup analyses | 12 months
  Pre-specified subgroup analyses will be conducted according to age, sex, education level, screening lifetime depression, employment type, work sector, years in employment, number of workers in the company, type of employment contract, work schedule, number of weekly hours worked and type of salary, as well as baseline measurements of anxiety and depression symptoms, risk level for depression, physical and mental quality of life, physical activity level, insomnia, social support, assertiveness, troubled relationship, and difficulties communicating or making decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Á Bellón, PhD, Principal Investigator — Andalusian Health Service
Locations (1):
- Juan Bellon Saameño, Málaga, Spain